CLINICAL TRIAL: NCT00693303
Title: Examining the Effectiveness of My Scrivener on Handwriting Legibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenandoah University (Other)
Responsible Party: Principal Investigator, Deborah Marr, Assistant Professor, Shenandoah University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-1125; #H133S070082 (Other: NIDRR)
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Results first posted 2009-08-25 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-06

CONDITIONS: Healthy Children
Keywords: single subject; quantitative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Handwriting Training using My Scrivener (Experimental): Subjects received 20 minutes of training per week which included writing letters and words with the My Scivener device.
  Interventions: Behavioral: Handwriting Training using My Scrivener

INTERVENTIONS:
Behavioral: Handwriting Training using My Scrivener — Subjects received 20 minutes of training per week which included writing letters and words with the My Scivener device.

SUMMARY:
The purpose of this study was to examine the changes in handwriting performance in elementary aged children who received handwriting training which included use of the My Scrivener stylus. Training on the My Scrivener stylus provided additional feedback to the children which is hypothesized to produce significant improvement.

DETAILED DESCRIPTION:
Once parental consent was given, students met individually with the PI or a trained occupational therapy graduate student in a private space at the Boys and Girls Club of the Northern Shenandoah Valley for a pre-test evaluation session. The evaluation consisted of the following:

1. Evaluation Tool of Children's Handwriting (ETCH; Amundson, 1995). This is a criterion-referenced tool measuring a child's legibility and speed in grades one through six. This measure is able to evaluate both manuscript and cursive handwriting; however, only the manuscript portion will be used as that will be the focus of the club's training. The ETCH asks the child to write letters and words in lower-case and upper-case, write numerals, perform near point and far point copying, write to dictation, and compose original sentences. Total time for the evaluation is 15-20 minutes.
2. Brief Assessment of Motor Function (BAMF: Parks, Cintas, Chaffin, & Gerber, 2007). This is a criterion referenced tool that can identify gross, fine, and oral motor performance in as little as 10 minutes. For this particular study, only the Fine Motor Scale of the BAMF will be used. Data from this tool will be used to categorize subjects for between group comparisons.
3. The Developmental Test of Visual Motor Integration (VMI: Beery, 1998). This gold-standard tool measures a child's visual motor performance by asking them to copy geometric shapes ranging from the very simple to the very complex. Data from this tool will be used to categorize subjects for between group comparisons.

Once all children were evaluated, twice weekly Handwriting Camp sessions were held. During these small group sessions lasting approximately 30 minutes each, 4 children at a time received instruction from the Handwriting Without Tears Curriculum from either the PI or trained OT graduate students and 20 minutes of supervised practice time on the My Scrivener equipment to reinforce the letter writing instruction for that day.

The Handwriting Camp sessions lasted for approximately 8 weeks.

At the conclusion of the camp, the pre-tests were re-administered as well as an open-ended question interview was conducted on how well the child enjoyed using the device.

ELIGIBILITY:
Inclusion Criteria:

* The subjects were any child enrolled in the summer program at the Boys and Girls Club of the Northern Shenandoah Valley entering grades 1 to 6 in Fall 2008 whose parents give consent.

Exclusion Criteria:

* None

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Marr, ScD, Principal Investigator — Shenandoah University
Locations (1):
- Boys and Girls Club of the Northern Shenandoah Valley, Winchester, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- My Scrivener Training: Subjects practiced writing letters and words for 20 minutes two times per week using the My Scrivenor device.
Period: Overall Study
Arm/Group | My Scrivener Training
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- My Scrivener Training: Children received My Scrivenor training
Arm/Group | My Scrivener Training
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 21
Evaluation Tool of Children's Handwriting [Mean (Standard Deviation); unit: Mean percent of legible letters, & words] — This criterion-referenced tool measures legibility and speed in grades one through six. The ETCH asks the child to write letters and words in lower-case and upper-case, write numerals, perform near point and far point copying, write to dictation, and compose original sentences.
  Mean percent of legible letters, & words | 95 (9.9)

OUTCOME MEASURES:

1. Primary Outcome: Evaluation Tool of Children's Handwriting
Description: This criterion-referenced tool measures a child's legibility and speed in grades one through six. The child writes letters and words, numerals, performs near point and far point copying, writes to dictation, and composes a sentence.
Time Frame: 8 weeks from start of training
Measure: Mean (Standard Deviation); unit: percent of legible letters
Arm/Group | My Scrivener Training
Number analyzed (Participants) | 21
percent of legible letters | 96 (6.9)
Statistical Analysis 1: Comparison: My Scrivener Training; Test type: Superiority or Other; p = .27, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | My Scrivener Training
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No